CLINICAL TRIAL: NCT02608684
Title: A Phase II Study of Pembrolizumab With Cisplatin and Gemcitabine Treatment in Patients With Recurrent Platinum-resistant Ovarian Cancer
Brief Title: A Study of Pembrolizumab With Standard Treatment in Patients With Recurrent Platinum-resistant Ovarian Cancer
Acronym: PemCiGem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Bobbie Jo Rimel, MD, Associate Professor, Obstetrics and Gynecology, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015-13-Walsh-PemCiGem
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer
Keywords: immunotherapy; platinum-resistant ovarian cancer; immune checkpoint inhibitors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pembrolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cisplatin+Gemcitabine+Pembrolizumab (Experimental): 2 cycles of 750mg gemcitabine and 30mg cisplatin chemotherapy (standard of care) followed by 4 cycles of gemcitabine and cisplatin combined with pembrolizumab in 21-day treatment cycles followed by single-agent pembrolizumab maintenance therapy for up to 2 years of treatment (6 cycles combination treatment + 28 cycles maintenance).
  Gemcitabine 750 mg/m2 every 3 weeks (Q3W) x 6 cycles IV infusion
  -Day 1 and Day 8 of each 3 week cycle Standard of care
  Cisplatin 30 mg/m2 Q3W x 6 cycles IV infusion
  -Day 1 and Day 8 of each 3 week cycle after gemcitabine Standard of care
  Pembrolizumab 200 mg Q3W starting with cycle 3 IV infusion
  -Day 1 of each 3 week cycle after gemcitabine and cisplatin Experimental
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab IV solution
  Other Names: Keytruda; MK-3475
Drug: Gemcitabine — Gemcitabine IV solution
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin IV solution
  Other Names: Platinol

SUMMARY:
To evaluate the efficacy and safety of anti-PD-1 antibody MK-3475 (pembrolizumab) in combination with gemcitabine and cisplatin chemotherapy in women with recurrent platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase II trial to evaluate the efficacy and safety of anti-PD-1 antibody MK-3475 (pembrolizumab) in combination with standard of care gemcitabine and cisplatin chemotherapy in women with recurrent platinum-resistant ovarian cancer (encompasses ovarian, peritoneal and fallopian tube cancer). Subjects will receive 2 cycles of gemcitabine and cisplatin chemotherapy followed by 4 cycles of gemcitabine and cisplatin combined with pembrolizumab in 21-day treatment cycles. Subjects will continue to receive single-agent pembrolizumab every 21 days as maintenance therapy for up to 2 year until progression or the subject meets withdrawal criteria. Tumor imaging with CT scan will occur at baseline and every 6 weeks (after each second cycle) during chemotherapy treatment and every 9 weeks thereafter. The primary endpoint is efficacy as defined overall response rate by Response Evaluation Criteria in Solid Tumors (RECIST v.1.1). Secondary endpoints for efficacy include progression free survival at 6 and 12 months, time to progression, duration of response and overall survival. Safety and tolerability of the regimen will be determined by assessing the frequency and intensity of adverse events as defined by the Common Terminology Criteria for Adverse Events (CTCAE v.4). Quality of life will be measured using the European Organization for Research and Treatment of Cancer quality of life questionnaire (QLQ-C30).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/ for the trial.
* Be at least 18 years of age on day of signing informed consent.
* Have histologically confirmed diagnosis of recurrent epithelial ovarian, peritoneal or fallopian tube carcinoma that has progressed within 6 months of prior cytotoxic chemotherapy. Histologic confirmation of the primary tumor by review of the pathology report is required. Patients must have had at least one prior platinum-based chemotherapeutic regimen. Initial treatment may have been administered as an intraperitoneal, intravenous or dose-dense regimen. Progression within 6 months of a non-platinum containing regimen is eligible if the patient is considered platinum-resistant to the last platinum-containing regimen. Patients who have received prior cisplatin and gemcitabine treatment are eligible to participate.
* Have measurable disease based on RECIST 1.1
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function, all screening labs should be performed within 28 days of treatment initiation.
* Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Patients who have had prior hysterectomy and/or bilateral oophorectomy are not required to have a pregnancy test.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.

Note: If subject received major surgery including (curative or palliative surgery), they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Note: Patients who have hypertension as an adverse event related to prior angiogenesis targeted therapy may be allowed if ≤ Grade 2 and considered by investigator to be well-controlled on anti-hypertensive agents.

* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the trial, starting with screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or positive serum test for HIV as per testing at screening
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) as per test at screening
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bobbie J Rimel, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin+Gemcitabine+Pembrolizumab: 2 cycles of 750mg gemcitabine and 30mg cisplatin chemotherapy (standard of care) followed by 4 cycles of gemcitabine and cisplatin combined with pembrolizumab in 21-day treatment cycles followed by single-agent pembrolizumab maintenance therapy for up to 2 years of treatment (6 cycles combination treatment + 28 cycles maintenance).
  Gemcitabine 750 mg/m2 every 3 weeks (Q3W) x 6 cycles IV infusion
  -Day 1 and Day 8 of each 3 week cycle Standard of care
  Cisplatin 30 mg/m2 Q3W x 6 cycles IV infusion
  -Day 1 and Day 8 of each 3 week cycle after gemcitabine Standard of care
  Pembrolizumab 200 mg Q3W starting with cycle 3 IV infusion
  -Day 1 of each 3 week cycle after gemcitabine and cisplatin Experimental
  Pembrolizumab: Pembrolizumab IV solution
  Gemcitabine: Gemcitabine IV solution
  Cisplatin: Cisplatin IV solution
Period: Overall Study
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Started | 21
Completed | 18
Not Completed | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ashkenazi Jewish - 0% | 14
  Ashkenazi Jewish - 100% | 3
  Ashkenazi Jewish - Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Defined as complete or partial response per RECIST 1.1 criteria with assessment every 6 weeks during first 6 cycles of therapy and every 9 weeks thereafter. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
Participants
  Complete Response | 1
  Partial Response | 10
  Stable Disease | 5
  Progressive Disease | 2

2. Secondary Outcome: Overall Response Rate by iRECIST
Description: Per Immune Response Evaluation Criteria In Solid Tumors Criteria (iRECIST) for target lesions and assessed by CT or MRI, where the threshold is reset if RECIST 1.1 progression is followed at the next assessment by tumor shrinkage: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0
  Progressive Disease | 12
  Not applicable | 6

3. Secondary Outcome: Progression-free Survival (PFS) at 6 Months and at 12 Months
Description: Percentage of patients who have not progressed at 6 and 12 months with progression-free survival calculated from the start of treatment to the date of progression or death from any cause. Progression is measured by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Progressive Disease (PD), At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest sum on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression.
Time Frame: 6 months and 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
percentage of participants
  PFS rate at 6 months | 50.00 [25.93 to 70.05]
  PFS rate at 12 months | 5.56 [0.37 to 22.42]

4. Secondary Outcome: Time to Progression
Description: Calculated in months from the start of treatment to disease progression as defined by Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI: Progressive Disease (PD), At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest sum on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
months | 6.25 [3.78 to 7.7]

5. Secondary Outcome: Duration of Response
Description: Calculated in months as time from documentation of tumor response to disease progression
Time Frame: Up to 2 years
Population: Among subjects who had a partial or complete response to treatment
Measure: Median (Full Range); unit: months
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 11
months | 3.75 [0.86 to 25.1]

6. Secondary Outcome: Overall Survival (OS)
Description: Calculated in months from the start of treatment to the date of death from any cause
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
months | 17.75 [7.47 to 32.24]

7. Secondary Outcome: Frequency and Intensity of Adverse Events (CTCAE v.4), Deemed at Least Possibly Related to Study Participation
Description: As measured at each visit, during safety follow up (30 days after discontinuation of treatment) and during follow up (every nine weeks after discontinuation). Adverse events graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4, with events graded from 1 to 5, where a higher grade reflects greater symptom severity.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
Number analyzed (Participants) | 18
Participants
  Alanine aminotrasferase increased, Grade 1 | 1
  Alanine aminotransferase increased, Grade 2 | 1
  Alanine aminotransferase increased, Grade 3 | 1
  Alopecia, Grade 1 | 1
  Anemia, Grade 2 | 3
  Anemia, Grade 3 | 3
  Anorexia, Grade 1 | 2
  Anorexia, Grade 2 | 2
  Aspartate aminotransferase increased, Grade 1 | 1
  Aspartate aminotransferase increased, Grade 2 | 1
  Aspartate aminotransferase increased, Grade 3 | 1
  Bilateral tinnitus, Grade 1 | 1
  Chills, Grade 1 | 1
  Dehydration, Grade 1 | 1
  Dehydration, Grade 3 | 1
  Diarrhea, Grade 1 | 3
  Diarrhea, Grade 3 | 1
  Edema limbs, Grade 2 | 1
  Edema limbs, Grade 3 | 1
  Fatigue, Grade 1 | 7
  Fatigue, Grade 2 | 2
  Fatigue, Grade 3 | 1
  Febrile neutropenia, Grade 3 | 1
  Headache, Grade 1 | 1
  Hearing impaired, Grade 1 | 1
  Hemolysis, Grade 3 | 1
  Hyperthyroidism, Grade 1 | 1
  Hypophysitis, Grade 1 | 1
  Hypothyroidism, Grade 1 | 3
  Hypothyroidism, Grade 2 | 2
  Leukocytosis, Grade 2 | 1
  Localized edema, Grade 1 | 1
  Localized edema, Grade 2 | 1
  Lymphocyte count decreased, Grade 3 | 4
  Memory impaired, Grade 1 | 1
  Mucositis oral, Grade 2 | 1
  Nausea, Grade 1 | 6
  Nausea, Grade 2 | 8
  Nausea, Grade 3 | 4
  Neutrophil count decreased, Grade 1 | 1
  Neutrophil count decreased, Grade 2 | 5
  Neutrophil count decreased, Grade 3 | 11
  Neutrophil count decreased, Grade 4 | 6
  Palpitations, Grade 2 | 1
  Peripheral sensory neuropathy, Grade 1 | 1
  Platelet count decreased, Grade 1 | 3
  Platelet count decreased, Grade 2 | 1
  Platelet count decreased, Grade 3 | 5
  Platelet count decreased, Grade 4 | 2
  Rash maculo-papular, Grade 1 | 1
  Skin hyperpigmentation, Grade 1 | 1
  Urine output decreased, Grade 3 | 1
  Vomiting, Grade 1 | 6
  Vomiting, Grade 2 | 7
  Vomiting, Grade 3 | 4
  Weight gain, Grade 1 | 1
  Weight gain, Grade 2 | 1
  White blood cell count decreased, Grade 3 | 6
  White blood cell count decreased, Grade 4 | 1

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cisplatin+Gemcitabine+Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 12/18
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin+Gemcitabine+Pembrolizumab (N=18)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypophysitis (Immune system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin+Gemcitabine+Pembrolizumab (N=18)
Abdominal pain (Gastrointestinal disorders) | 14 (23)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 5 (8)
Anxiety (Psychiatric disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 5 (7)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bilateral tinnitus (Ear and labyrinth disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 10 (14)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Dizziness (Nervous system disorders) | 2 (3)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (5)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Ear disorder (hot) (Ear and labyrinth disorders) | 1 (1)
Ear disorder (tingling) (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 13 (22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Heart murmur (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3)
Hypertension (Vascular disorders) | 7 (9)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (5)
Hypotension (Vascular disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 5 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileal obstruction (Gastrointestinal disorders) | 1 (1)
Infusion-related reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (8)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Localized edema (General disorders) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (8)
Malaise (General disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Multinodular goiter (Endocrine disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (27)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 13 (45)
Non-cardiac chest pain (General disorders) | 5 (7)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Papulopustular rash (Infections and infestations) | 1 (1)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5)
Platelet count decreased (Investigations) | 7 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash generalized (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (9)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thyroid nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Vaginal extrusion (Injury, poisoning and procedural complications) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 9 (29)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02608684/Prot_SAP_000.pdf